CLINICAL TRIAL: NCT02424721
Title: Prospective, Non-interventional, Multi-centre Clinical Study to Assess the Clinical Validity of the Heparin Binding Protein Assay to Assist in Evaluation of Patients With Suspected Infection Following Emergency Department Admission
Brief Title: Sepsis Assessment in Belgian Emergency Rooms
Acronym: SABER
Status: Terminated | Type: Observational
Why Stopped: Resource constraints at participating sites
Sponsor: Axis Shield Diagnostics Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: PEP-FMHBP-003
Record Dates: First submitted 2015-04-15; First posted 2015-04-23 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Sepsis; Shock, Septic; Severe Sepsis
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma - NaCitrate and LiHep

SUMMARY:
To validate the use of the Heparin Binding Protein (HBP) concentration to assist in the evaluation of patients admitting to the emergency department with suspected infection.

DETAILED DESCRIPTION:
Prospective, non-interventional, multi-centre clinical study to assess the clinical validity of the Heparin Binding Protein (HBP) assay to assist in evaluation of patients with suspected infection following emergency department admission.

Patients presenting to the emergency department with suspected infection will be enrolled to the study and have a blood sample taken.

The patients clinical data over a 72 hour period after enrolment will be recorded in the CRF. The enrolment sample will then be retrospectively measured for the HBP level and the power of the enrolment HBP level to predict subsequent clinical development over the following 72 hours will be assessed. Data analysis shall include Area Under Curve (AUC) from Receiver Operating Characteristics (ROC) plot against the patient's final clinical diagnosis as well as sensitivity and specificity of the HBP level to predict the final clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age,
* Suspected infection (temperature >38C or clinical evidence of infection),
* intention by clinician to start antibiotics

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the Emergency Department with suspected infection
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-05; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Validation of use of HBP in evaluation of patients with suspected infection | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Vincent, MD, Principal Investigator — Erasme University Hospital
Locations (4):
- Belgium (4):
  - Clinique St Anne St Remy, Anderlecht
  - Hopital Erasme, Brussels
  - Hopital Civil de Charleroi, Charleroi
  - CHU Tivoli, La Louvière